CLINICAL TRIAL: NCT04138550
Title: Exploring the Structural and Intermediary Social Determinants of Oral Health Among Egyptian Women: A Cross-Sectional Study
Brief Title: Structural and Intermediary Social Determinants of Oral Health Among Egyptian Women
Status: Not yet recruiting | Type: Observational
Sponsor: Misr International University (Other)
Responsible Party: Sponsor
Other Study IDs: PUB 1114003
Record Dates: First submitted 2019-10-21; First posted 2019-10-24 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-03

CONDITIONS: Oral Health
Keywords: Social determinants; Oral health; Women; Egypt

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Globally, there is substantial evidence indicating that low household income, lack of education, poor living conditions and inadequate psycho-social social support are potential risk factors for morbidity and premature death. Despite that, worldwide, there is scarcity in evidence on potential social determinants of oral health among different population groups.The study aims To identify the potential social determinants with an influence on oral health status of Egyptian women.

DETAILED DESCRIPTION:
Statement of problem

Globally, there is substantial evidence indicating that low household income, lack of education, poor living conditions and inadequate psychosocial social support are potential risk factors for morbidity and premature death. Despite that, worldwide, there is scarcity in evidence on potential social determinants of oral health among different population groups.

Aim of study

To identify the potential social determinants with an influence on oral health status of Egyptian women.

Materials and methods

A total of 300 Egyptian women in childbearing age (18-49 years) will be recruited from 4 Primary healthcare units in Qalyubia governorate in Egypt. Four trained investigators will conduct a face-to face interview with study participants to gather data on potential structural and intermediary social determinants of health using a questionnaire. The questionnaire is based upon The Commission on Social Determinants of Health (CSDH) conceptual framework which was set up by the World Health Organization in 2005. This tool includes questions on socioeconomic position, material factors and living conditions, psychosocial factors and behavioral factors. Caries experience and gingival health of participants will be determined using DMFT, DMFS and CPITN indices respectively.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian women in child bearing age (18-49 years) attending one of the governmental primary healthcare units.

Exclusion Criteria:

* Women who recently moved from one place of residence to another.
* Women attending the dental clinic at one of the primary health units selected for the survey.
* Pregnant Women.
* Completely Edentulous Women.
* Women with mental or psychological issues.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Egyptian women in child bearing age (18-49 years) attending one of the governmental primary healthcare units selected for the survey.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2027-12-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Social determinants | 11 months from enrollment
  Questionnaire Likert scale 1 - 5

SECONDARY OUTCOMES:
Caries Experience | 11 months from enrollment
  Decayed, Missed, Filled caries index: 0 - 32
Gingival/periodontal health | 11 months from enrollment
  Modified Community Periodontal Index: 0 - 4
Esthetics | 11 months from enrollment
  Number of unfilled upper spaces

CONTACTS AND LOCATIONS:
Overall Officials: Mahassen M. Farghaly, Professor, Study Director — MIU Vice President for Community Services and Environmental Affairs

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] Frieden TR. A framework for public health action: the health impact pyramid. Am J Public Health. 2010 Apr;100(4):590-5. doi: 10.2105/AJPH.2009.185652. Epub 2010 Feb 18. PMID 20167880
- [Background] Kwan S, Petersen PE. Oral health: equity and social determinants. In: Blas E, Sivansankara Kurup A, editors. Equity, social determinants and public health programmes. Geneva: World Health Organization, 2010; 159-76.
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Steele J, Shen J, Tsakos G, Fuller E, Morris S, Watt R, Guarnizo-Herreno C, Wildman J. The Interplay between socioeconomic inequalities and clinical oral health. J Dent Res. 2015 Jan;94(1):19-26. doi: 10.1177/0022034514553978. Epub 2014 Oct 24. PMID 25344336
- [Background] World Health Organization. A Conceptual Framework for Action on the Social Determinants of Health. 2010.
- [Background] Daly MC, Duncan GJ, McDonough P, Williams DR. Optimal indicators of socioeconomic status for health research. Am J Public Health. 2002 Jul;92(7):1151-7. doi: 10.2105/ajph.92.7.1151. PMID 12084700
- [Background] Melki IS, Beydoun HA, Khogali M, Tamim H, Yunis KA; National Collaborative Perinatal Neonatal Network (NCPNN). Household crowding index: a correlate of socioeconomic status and inter-pregnancy spacing in an urban setting. J Epidemiol Community Health. 2004 Jun;58(6):476-80. doi: 10.1136/jech.2003.012690. PMID 15143115
- [Background] Fatima A. Al-Ghadban. Evaluating the Face Validity of an Arabic-language Translation of a Food Security Questionnaire in Arabic-speaking Populations. THESIS 2012.
- [Background] Dahlem NW, Zimet GD, Walker RR. The Multidimensional Scale of Perceived Social Support: a confirmation study. J Clin Psychol. 1991 Nov;47(6):756-61. doi: 10.1002/1097-4679(199111)47:63.0.co;2-l. PMID 1757578
- [Background] Smith MS, Wallston KA, Smith CA. The development and validation of the Perceived Health Competence Scale. Health Educ Res. 1995 Mar;10(1):51-64. doi: 10.1093/her/10.1.51. PMID 10150421
- [Background] Acharya DR, Bell JS, Simkhada P, van Teijlingen ER, Regmi PR. Women's autonomy in household decision-making: a demographic study in Nepal. Reprod Health. 2010 Jul 15;7:15. doi: 10.1186/1742-4755-7-15. PMID 20630107
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Sanders AE 2007. Social Determinants of Oral Health: conditions linked to socioeconomic inequalities in oral health and in the Australian population. AIHW cat. no. POH 7. Canberra: Australian Institute of Health and Welfare (Population Oral Health Series No. 7).